CLINICAL TRIAL: NCT00699777
Title: A Randomized, Open-label, 2-period, Crossover Study to Assess the Bioequivalence of One 150 mg Risedronate Tablet Versus Two 75 mg Risedronate Tablets Administered as a Single Oral Dose in Healthy Male and Female Subjects
Brief Title: Assess Bioequivalence of One 150 mg Risedronate Tablet Versus Two 75 mg Risedronate Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2007141
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): One risedronate 150 mg tablet administered orally after an overnight (10 hour) fast, followed by a 4 hour post-dose fast
  Interventions: Drug: Risedronate
- 2 (Active Comparator): Two risedronate 75 mg tablets administered as a single oral dose after an overnight (10 hour) fast, followed by a 4 hour post-dose fast
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Risedronate — 1 risedronate 150 mg tablet administered orally
  Arms: 1
Drug: Risedronate — 2 risedronate 75 mg tablets administered as a single oral dose
  Arms: 2

SUMMARY:
This study is a randomized, open-label, crossover study to assess the bioequivalence of 1 risedronate 150 mg tablet versus 2 risedronate 75 mg tablets administered as a single oral dose. Approximately 320 subjects will be enrolled from 4 study centers in the U.S.

DETAILED DESCRIPTION:
The data to support the interchangeability of one risedronate 150 mg tablet versus two risedronate 75 mg tablets as monthly dose forms is primarily based on the similarity of in vitro dissolution and an in vivo study, which showed risedronate absorption is not dissolution rate limited. These results suggest that monthly dosing of risedronate may be accomplished by administration of either one risedronate 150 mg tablet or two risedronate 75 mg tablets. The purpose of this study is to provide additional clinical data to support the interchangeability of these 2 dose regimens.

ELIGIBILITY:
Inclusion Criteria:

* be in good general health based on medical history, physical examination, and laboratory evaluation
* have a body mass index (BMI) ≤ 32 kg/m2 at screening

Exclusion Criteria:

* has clinically significant uncontrolled cardiovascular, hepatic, renal, or thyroid disease
* has any disease or surgery known to alter normal GI structure or function
* has a creatinine clearance of < 60 mL/min, estimated by serum creatinine using the Cockcroft-Gault formula

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the bioequivalence of one risedronate 150 mg tablet versus two risedronate 75 mg tablets administered as a single oral dose. | 18-21 days

CONTACTS AND LOCATIONS:
Overall Officials: William S Aronstein, PhD/M/FACP, Study Director — Procter and Gamble
Locations (4):
- United States (4):
  - Research Site, Gainesville, Florida
  - Research Facility, Miramar, Florida
  - Research Facility, Austin, Texas
  - Research Facility, Dallas, Texas